CLINICAL TRIAL: NCT00569647
Title: Preoperative Anxiety in Pediatric Reconstructive Burn Patients: The Role of Virtual Reality Hypnosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: John E McCall MD PI, Shriners Hospital for Children
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 277444040
Record Dates: First submitted 2007-11-29; First posted 2007-12-07 (Estimated); Last update posted 2007-12-07 (Estimated); Status verified 2007-11

CONDITIONS: Anxiety
Keywords: preoperative anxiety; burn reconstruction
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- v (Experimental): Use of VRH headset
  Interventions: Device: Virtual Reality Hypnosis
- c (Placebo Comparator)
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Virtual Reality Hypnosis — Use of virtual reality headset to induce hypnotic state
  Arms: v
Device: Placebo — no use of device
  Arms: c

SUMMARY:
Children with burns often require repeated reconstructive surgeries. These children tend to develop high levels of anxiety before coming to the operating room. Preoperative sedation, while somewhat effective in relieving this anxiety, has a number of side effects. The researchers hypothesized that preoperative anxiety could be effectively reduced by the utilization of a device which induces a relaxing hypnotic state through emmersion in a virtual reality environment.

DETAILED DESCRIPTION:
The virtual reality environment is created by a Virtual Reality Hypnosis (VRH) device. The patient wears a headset which contains video and audio display. A twenty minute program is viewed, which guides the patient into a relaxed state via soothing audio and video input.

ELIGIBILITY:
Inclusion Criteria:

* Child presenting for reconstructive burn surgery

Exclusion Criteria:

* Visual or auditory difficulties

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2005-11; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
anxiety reduction | preoperatively

CONTACTS AND LOCATIONS:
Overall Officials: John E McCall, MD, Principal Investigator — University of Cincinnati